CLINICAL TRIAL: NCT04471142
Title: Effectiveness of Compressive Bandage Use in Post-Treatment Seroma Prevention Breast Cancer Surgery
Brief Title: Effectiveness of Compressive Bandage Use in Seroma Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Principal Investigator, Erica Alves Nogueira Fabro, INCA Effectiveness Seroma Prevention, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Instituto Nacional do Câncer
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Seroma
Keywords: physiotherapy; seroma; breast cancer; taping
MeSH Terms: conditions — Seroma; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients undergoing mastectomy will be evaluated for eligibility criteria after the first dressing, those considered eligible will be randomized to the intervention or control group. 27 blocks will be available containing 10 envelopes where 05 will contain a code that allocates the patients in group A and 05 in group B. Group A: intervention group with preventive application of compressive bandage in addition to the suction drain (routine adopted in the institution). The bandage will be applied on the day of discharge after the first dressing, withdrawal and new bandage applied on the fourth day and permanently removed on the seventh day when they will be reevaluated. Group B: control group. Patient will follow the routine of the institution only with the suction drain.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A (Experimental): Intervention group with preventive application of compressive bandages in addition to suction drain (routine adopted at the institution).
  Interventions: Device: neuromuscular bandage
- Group B (No Intervention): Group control. The patient will follow the institution's routine with only the suction drain.

INTERVENTIONS:
Device: neuromuscular bandage — After the dressing is performed by the nursing team with a sterile gauze covering over the region of the healing points, the 7 cm wide Vitaltape® neuromuscular bandage will be applied. For the application of the bandage, maximum stretching will be performed over the region of the plastron and finished with the two ends, from two to three centimeters, without stretching. As many bundles of bandages as necessary will be applied according to the patient's body characteristics.
  Other Names: compressive taping; compressiva bandage
  Arms: Group A

SUMMARY:
INTRODUCTION: Seroma is the most common complication after surgical treatment for breast cancer. It is the abnormal accumulation of serous fluid that develops under skin flaps and may be associated with necrosis, dehiscence, sepsis, and shoulder dysfunction. The therapeutic bandage has been inserted in clinical practice because it is similar to the elasticity of the skin and is able to help the circulatory and lymphatic system, reduce pain and local swelling, and may have benefits for prevention and treatment of seroma when applied compressively. . OBJECTIVE: To evaluate the effectiveness of compressive bandage in preventing seroma. METHODOLOGY: Randomized study of women over 18 years who underwent mastectomy at HCIII / INCA. Eligible patients will be allocated to the intervention and control groups by lot (270 envelopes, 135 patients per group). The intervention group, in addition to the use of the drain, will be submitted to the compression bandage on the day of hospital discharge and will be reevaluated on the seventh day. The control group will follow the institutional routine, using only the drain. The incidence and volume of the seroma, as well as the length of stay of the drain will be evaluated after 30 days through the medical record. Symptoms and skin changes resulting from the use of the bandage will be evaluated through a specific form. ANALYSIS: Descriptive analysis will be by measures of central tendency, dispersion and frequency distribution. Outcome assessment will be performed by odds ratio (for categorical variables) and by mean difference (Student's t-test), considering a 95% confidence interval. To control the confounding variables, multiple logistic regression (categorical outcome) and multiple linear regression (continuous outcome) will be performed by the Stepwise Forward method, including variables with p <0.20.

DETAILED DESCRIPTION:
This is a randomized clinical trial with women undergoing surgical treatment for breast cancer at Cancer Hospital III / INCA. All patients undergoing mastectomy will be evaluated for eligibility criteria after the first dressing in the hospital, those considered eligible will be informed about the study and no obligation to participate through free and informed consent. Upon acceptance, patients will be randomized to the intervention or control group, which will be performed by lot at the time the patient enters the study. 27 blocks will be available containing 10 envelopes where 05 will contain a code that allocates the patients in group A and 05 in group B. This choice was chosen to avoid influences of the therapist or patient's preference over the intervention. The patients will be oriented in relation to the group they are inserted and what monitoring will be performed while the patient is under the care of the dressing. All evaluations, intervention and data collection will be performed by trained professionals qualified for this purpose. Group A: intervention group with preventive application of compressive bandage in addition to the suction drain (routine adopted in the institution). Patients allocated to this group on the day of the first dressing, before hospital discharge, according to the institutional routine, are instructed by the nursing staff to wash the plastron region with cold, boiled filtered water and to return within one week at the outpatient clinic. The bandage will be applied on the day of discharge after the first dressing, withdrawal and new bandage applied on the fourth day and definitive removal on the seventh day when it will be scheduled for return in nursing care. Should any complications occur due to the use of the bandage, the patients will be advised to remove the material at home and will be suspended from the research protocol. At the end of the seven days, the patients will be reevaluated. Prior to the application of the bandage will be made the antisepsis of the skin and placement of the transparent and sterile film dressing over the region of the scar points to protect the scar. The 5 cm wide Vitaltape® neuromuscular bandage will be used with maximum stretching over the plastron region and finished with two ends of two to three centimeters without stretching. As many bundles of bandages as necessary will be applied according to the patient's body characteristics. All applications will be performed by the same physical therapist. Group B: control group. The patient will follow the institution's routine only with the suction drain. All patients will be instructed to do the same care with the suction drain according to the institutional routine.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over
* underwent mastectomy assurgical treatment for breast cancer.

Exclusion Criteria:

* bilateral breast cancer;
* patient undergoing neoadjuvant radiotherapy;
* infection in the surgical wound or hematoma;
* autoimmune disease reporting (dermatomyositis, hidradenitis suppurativa, nephropathy, lupus erythematosus, morphea, psoriasis, pemphigus vulgaris, scleroderma);
* patients with difficulties in understanding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2021-11-08 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Seroma Incidence | 30 days
  the presence of assessed local fluctuation will be considered seroma by the nursing team during dressing care, with indication of puncture aspiration to resolve the condition, regardless of the volume drained.
Seroma volume | 30 days
  the total volume drained and the number of aspirations will be considered necessary until resolution of the picture.
Permanence time with the Suction Drain | 15 days
  The permanence time (in days) will be checked with the suction drain, as reported by the dressing team.

SECONDARY OUTCOMES:
Safety of the use of the compressive bandage in mastectomized women | 7 days
  The dermal changes will be evaluated at the location of the bandage application of the 135 participants in the intervention group, such as discoloration, increased local temperature, skin peeling, presence of a wound and formation of bullous lesions at the site of the application of the neuromuscular bandage, graded in light, moderate or severe, according to the severity of the change, from a semi-structured questionnaire.
To assess the tolerance reported by the patient to the use of compressive taping | 7 days
  The symptoms of pain, itching, burning, discomfort, tightness, increased fluctuation of the seroma at the site of application of the bandage of the 135 participants will be evaluated. The symptoms will be graded according to the Visual Numeric Scale (0-10), where 0 will be considered no sensation and 10 unbearable sensation with the use of the bandage.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Fabro, Master, Principal Investigator — INCA - Brazil
Locations (1):
- Erica Alves Nogueira Fabro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Fabro EAN, Costa RM, Fernandes MC, Ximenes MA, Nogueira DA, Soares NB, Thuler LCS, Bergmann A. Seroma incidence and risk factors in women undergoing mastectomies as surgical breast cancer treatment. Support Care Cancer. 2024 Sep 25;32(10):688. doi: 10.1007/s00520-024-08881-w. PMID 39322817
- [Derived] Fernandes MC, Fabro EAN, Ximenes MA, Costa RMM, Soares NB, Aguiar SS, Thuler LCS, Bergmann A. Compressive taping to prevent postmastectomy seroma: patient adherence and satisfaction. BMJ Support Palliat Care. 2024 May 17:spcare-2024-004912. doi: 10.1136/spcare-2024-004912. Online ahead of print. PMID 38760081